CLINICAL TRIAL: NCT04694105
Title: Peri-neural Dexmedetomidine Versus Dexamethasone as an Adjuvant to Bupivacaine Single Injection in Ultrasoundguided Supraclavicular Brachial Plexus Block for Arteriovenous Fistula: A Randomized Controlled Study
Brief Title: Peri-neural Dexmedetomidine Versus Dexamethasone for Supraaclavicular Block Adjuvant to Bupivacaine Supraclavicular Brachial Plexus Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, mahmoud salem soliman, Head of intensive care unit at new kaser al ainy teaching hospital , lecterur of anaesthesia and intensive care cairo universty, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: regional block adjuvants
Record Dates: First submitted 2020-12-18; First posted 2021-01-05 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Brachial Plexus Block
Keywords: dexmedetomidine; dexamethasone
MeSH Terms: interventions — Dexmedetomidine; Dexamethasone; Sodium Chloride; Saline Solution

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Care Provider
Masking Description: double blind both anesthetist and patient not aware about type of local anesthesia
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- dexmedetomidine (Active Comparator): Bupivacaine 30 ml 0.25% was combined with 50 microgram (0.5 ml) peri-neural dexmedetomidine plus 1.5 ml normal saline
  Interventions: Drug: Dexmedetomidine injection
- dexamethasone (Active Comparator): Bupivacaine 30 ml 0.25% was combined with 4 mg peri neural dexamethasone (2 ml)
  Interventions: Drug: Dexamethasone
- control group (Placebo Comparator): Bupivacaine 30 ml 0.25% was combined with 2 ml normal saline
  Interventions: Drug: saline

INTERVENTIONS:
Drug: Dexmedetomidine injection — perineural injection of Bupivacaine 30 ml 0.25% combined with 50 microgram (0.5 ml) peri-neural dexmedetomidine plus 1.5 ml normal saline
  Other Names: precedex
  Arms: dexmedetomidine
Drug: Dexamethasone — perineural injection of Bupivacaine 30 ml 0.25% combined with 4 mg peri neural dexamethasone (2 ml)
  Other Names: decadrone
  Arms: dexamethasone
Drug: saline — perineural injection of Bupivacaine 30 ml 0.25% combined with 2 ml normal saline
  Other Names: normal saline
  Arms: control group

SUMMARY:
to assessthe impact of addition of Dexmedetomidine or Dexamethasone to Bupivacaine, on Duration of analgesia (time in hours to the first report of postoperative pain )at the surgical site

DETAILED DESCRIPTION:
This randomized, controlled double blinded study included 42 adult patients undergoing arteriovenous fistula surgery. Ultrasound-guided supraclavicular brachial plexus block was initiated after placement of full monitoring . Supraclavicular brachial plexus block was achieved with the use of total volume 32 ml of anesthetic drugs in all patients. Bupivacaine 30 ml 0.25% was combined with 2 ml normal saline (control group A, n=14), Bupivacaine 30 ml 0.25% was combined with 50 microgram (0.5 ml) peri-neural dexmedetomidine plus 1.5 ml normal saline ( dexmedetomidine group B ,n=14), or Bupivacaine 30 ml 0.25% was combined with 4 mg peri neural dexamethasone (2 ml) ( dexamethasone group C, n=14).The onset and duration of sensory and motor blocks, the time to first request to postoperative rescue analgesic, Richmond Agitation-Sedation Score, hemodynamic data, visual analogue pain scores, were reported at predetermined time assessment points. Postoperative rescue intravenous fentanyl consumption over 24 hours and complications occurred were recorded.

ELIGIBILITY:
Inclusion Criteria:

* All the patients included in the study aged 18 to 60 years old were on chronic hemodialysis and they had a hemodialysis session one day before the block performance

Exclusion Criteria:

* Neurological, neuromuscular, psychiatric disorders, hepatic, respiratory, or cardiac diseases; coagulation disorders; infection at the block injection site; patients with a body mass index more than 35; or patients who refused the procedure

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-01-12 (Actual)

PRIMARY OUTCOMES:
Duration of analgesia | "UP to 4 hours post operative"
  (time in hours to the first report of postoperative pain at the surgical site, administered of opioid when VAS score was>4).

SECONDARY OUTCOMES:
Pain scores. | "at 8 and 24 hours post operative"
  Severity of pain at the surgical site (VAS) score

CONTACTS AND LOCATIONS:
Overall Officials: Tarek A Radwan, MD, Study Director — Cairo University
Locations (1):
- Kasr Alini Univeristy Hospital, Cairo, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kulenkampff D. BRACHIAL PLEXUS ANAESTHESIA: ITS INDICATIONS, TECHNIQUE, AND DANGERS. Ann Surg. 1928 Jun;87(6):883-91. doi: 10.1097/00000658-192806000-00015. No abstract available. PMID 17865904
- [Result] Neal JM. Ultrasound-Guided Regional Anesthesia and Patient Safety: Update of an Evidence-Based Analysis. Reg Anesth Pain Med. 2016 Mar-Apr;41(2):195-204. doi: 10.1097/AAP.0000000000000295. PMID 26695877
- [Result] Ji F, Li Z, Nguyen H, Young N, Shi P, Fleming N, Liu H. Perioperative dexmedetomidine improves outcomes of cardiac surgery. Circulation. 2013 Apr 16;127(15):1576-84. doi: 10.1161/CIRCULATIONAHA.112.000936. Epub 2013 Mar 19. PMID 23513068